CLINICAL TRIAL: NCT06134973
Title: A Prospective Study on the Application of Liquid Biopsy in the Surveillance of High-risk Population of Hepatocellular Carcionoma.
Brief Title: A Prospective Study on the Application of Liquid Biopsy in the Surveillance of High-risk Population of HCC.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Third Central Hospital (Other)
Collaborators: BGI, China (Other)
Responsible Party: Sponsor
Other Study IDs: Fangwang03
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Liquid biopsy; ultrasonic testing
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nodular group: nodules less than 2 cm in diameter
  Interventions: Diagnostic Test: ultrasonic testing
- Macronodular group: nodules between 2-3 cm in diameter
  Interventions: Diagnostic Test: ultrasonic testing

INTERVENTIONS:
Diagnostic Test: ultrasonic testing — ultrasonic testing

SUMMARY:
Liquid biopsy technology based on high-throughput sequencing can detect trace signals in the early stage of cancer in plasma free DNA, so it has become a new technology suitable for tumor diagnosis and screening.Relying on the key discipline of digestive liver disease in our hospital, this project cooperated with BGI to jointly carry out a prospective study on the application of liquid biopsy in the monitoring of population at risk of liver cancer by taking advantage of its technical advantages in next-generation sequencing, so as to provide an innovative way for the prevention and treatment of Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
Hepatocellular Carcinoma (HCC)is one of the cancers with high morbidity and mortality in the world , and the incidence of liver cancer in China is particularly serious. In 2020, there will be 410,000 new cases of liver cancer in China, accounting for 42.5% of the world. There were 391,000 deaths, ranking fifth in the incidence of malignant tumors and second in the fatality rate . Most patients with primary liver cancer have insidious onset and have reached the middle and late stage when diagnosed. At this time, the treatment of liver cancer is few, the prognosis is poor, and the mortality is high.Early detection and treatment are of great significance to improve the survival rate of patients with liver cancer, and the 5-year survival rate after early liver cancer (BCLC stage 0/A) can reach more than 60%. However, the diagnosis rate of early liver cancer in China is only 30%. In other countries, early diagnosis rates can be increased to more than 60% by monitoring high-risk populations. It can be seen that close monitoring of the pre-cancer stage is the key to early diagnosis and early treatment of HCC.

Identifying people at high risk for cancer development is the premise of cancer Surveillance and the biggest difference from conducting tumor Screening in the general population. Compared with many other common cancers, Targets for liquid biopsies come in many forms, including genetics-based tests for gene mutations, and epigenetic-based tests for methylation. Since no specific gene mutation events directly related to cancerization have been found in liver cancer, the effect of searching for biomarkers along this route is limited. Therefore, detecting early liver cancer from the epigenetic level has become another way worth exploring.

In the epigenetic mechanism, DNA methylation is an important gene regulation mode, which is closely related to the occurrence and development of tumors. More importantly, abnormal methylation of cancer-related genes often occurs in the early stage of cancer development, so DNA methylation signals are considered as potential markers for early tumor screening [14]. In addition, methylation modification is tissue-specific in different tumors and can even be used to locate the primary tissue of cancer, which is an ideal molecular marker for tumor early screening [15]. Therefore, ctDNA, which carries tumor cell-specific methylation information, can be used as a target for liquid biopsy of liver cancer, providing an innovative path for early diagnosis of HCC develops gradually on the basis of clear causes, such as typical hepatitis, cirrhosis to liver cancer "three steps". These characteristics determine the target population for early diagnosis of HCC, which can be found in the medical treatment of various chronic liver diseases. Making full use of these precancerous risk factors and identifying high-risk groups of liver cancer as surveillance objects will help improve the detection rate of cancer and obtain a better benefit-cost ratio.

Intrahepatic nodules are the disorder of hepatic trabecular arrangement caused by fibrous tissue hyperplasia. Their formation indicates the progression of liver injury and is also an important stage of precancerous lesions. Pathologically, nodules can be divided into stages such as regenerated nodules, low grade and high grade atypical hyperplasia, and adenoma according to their proximity to cancer, but the standards and terminology are still difficult to be unified, and pathological diagnosis requires obtaining samples through liver puncture, which is not widely used in clinical practice. In this case, the size of the intrahepatic nodules detected by ultrasound becomes an important basis for liver cancer risk stratification. Taking the current guidelines for diagnosis and treatment of liver cancer in China as an example, whether the nodule diameter is greater than 2 cm is the main basis for classification and diagnosis: for nodules less than 2 cm, at least two imaging evidences are required to confirm liver cancer; For nodules larger than 2 cm, only one item is needed. In addition, stratified analysis based on the size of intrahepatic nodules is also a framework for objective evaluation of the role of tumor markers. Alpha-fetoprotein (AFP), a traditional serum marker for hepatocellular carcinoma, has a sensitivity of 72-87% in advanced hepatocellular carcinoma. But for early-stage liver cancer smaller than 2 cm, its sensitivity is only 30-50%.

In view of the shortcomings of traditional serological markers with few types and low specificity, many important advances have been made in the application of molecular detection techniques based on omics to cancer diagnosis and screening. The liquid biopsy technology based on high throughput sequencing can detect specific abnormal signals in a small amount of Circulating Tumor DNA (ctDNA) in human peripheral blood, thus promoting the technological innovation of tumor early screening.

Targets for liquid biopsies come in many forms, including genetics-based tests for gene mutations, and epigenetic-based tests for methylation. Since no specific gene mutation events directly related to cancerization have been found in liver cancer, the effect of searching for biomarkers along this route is limited. Therefore, detecting early liver cancer from the epigenetic level has become another way worth exploring.

In the epigenetic mechanism, DNA methylation is an important gene regulation mode, which is closely related to the occurrence and development of tumors. More importantly, abnormal methylation of cancer-related genes often occurs in the early stage of cancer development, so DNA methylation signals are considered as potential markers for early tumor screening . In addition, methylation modification is tissue-specific in different tumors and can even be used to locate the primary tissue of cancer, which is an ideal molecular marker for tumor early screening . Therefore, ctDNA, which carries tumor cell-specific methylation information, can be used as a target for liquid biopsy of liver cancer, providing an innovative path for early diagnosis of HCC.

Although liquid biopsy shows promising application in the early diagnosis of HCC, most results are based on retrospective studies. According to the steps of marker research and development, future and multi-center studies are needed to verify it. In this project, we will rely on the team and work foundation of the key discipline of digestion (Liver disease), and cooperate with BGI Shenzhen BGI Medical Laboratory to carry out liquid biopsy based on methylation, and evaluate its feasibility for liver cancer monitoring through prospective studies. Promote the realization of early detection, diagnosis and treatment of HCC.

The risk assessment model of liver cancer was established to identify the high-risk groups of liver cancer. A prospective cohort study was conducted to evaluate the predictive ability of liquid biopsy technology for liver cancer occurrence, and to verify the performance and application prospects of this novel genetic detection technology in liver cancer monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as chronic liver disease, including but not limited to chronic hepatitis B, chronic hepatitis C, fatty liver;
2. Intrahepatic nodules detectable by ultrasound;
3. Unlimited number of nodules;
4. The patient has signed an informed consent form.

Exclusion Criteria:

1. Previously diagnosed malignant tumors；
2. Patients who are unable to cooperate with venous blood sampling；
3. According to the judgment of the investigator, the participants are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment criteria: All patients who were admitted to our hospital over 18 years old and found intrahepatic nodules by abdominal ultrasound and consented to join the prospective cohort study of intrahepatic nodules monitoring. Enrolled patients were grouped according to the maximum diameter of nodules in the live and were divided into nodular group (diameter less than 2 cm) and macronodular group (diameter 2-3 cm).
  Outcome events: Intrahepatic nodules were diagnosed as cancerous nodules. Follow-up: Patients who found intrahepatic nodules but were not confirmed by imaging or pathology were followed up every 2-3 months with imaging combined with serum AFP levels until the outcome events were observed.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The establishment of risk assessment model | 6-12 months
  The risk assessment model of liver cancer was established to identify the high-risk groups of HCC.
Application prospect of liquid biopsy technique in monitoring HCC in high risk population | 12-24 months
  To evaluate the potential application of liquid biopsy techniques for liver cancer surveillance in high-risk populations through a prospective cohort

CONTACTS AND LOCATIONS:
Overall Officials: Fengmei Wang, PhD, Principal Investigator — Tianjin Third Central Hospital
Locations (1):
- 王芳, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No